CLINICAL TRIAL: NCT01550354
Title: Comparison Among Propofol, Alfentanil and Rocuronium as Adjunct to Sevoflurane Anesthesia for Endotracheal Intubation in Children With Frenectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 4-2011-0824
Record Dates: First submitted 2012-02-22; First posted 2012-03-12 (Estimated); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Ankyloglossia
MeSH Terms: conditions — Ankyloglossia

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Propofol group (Active Comparator): Intravenous administration of propofol 2 mg/kg before intubation
  Interventions: Drug: administration of propofol
- Alfentanil group (Active Comparator): Intravenous administration of alfentanil 14 μg/kg before intubation
  Interventions: Drug: administration of alfentanil
- Rocuronium group (Active Comparator): Intravenous administration of rocuronium 0.3 mg/kg before intubation
  Interventions: Drug: administration of rocuronium

INTERVENTIONS:
Drug: administration of propofol — intravenous administration of propofol 2 mg/kg before intubation
  Arms: Propofol group
Drug: administration of alfentanil — intravenous administration of alfentanil 14 μg/kg before intubation
  Arms: Alfentanil group
Drug: administration of rocuronium — Intravenous administration of rocuronium 0.3 mg/kg before intubation
  Arms: Rocuronium group

SUMMARY:
Several methods have been demonstrated to improve intubating conditions during sevoflurane induction in children. These include opioids, propofol, and addition of neuromuscular blocking agents in pediatric patients. But the study about the comparison of these agents has been uncommon. Frenectomy is common procedure to treat ankyloglossia. It is a short procedure performed under general anesthesia. The investigators aimed to compare intubating conditions among children with propofol, alfentanil or rocuronium after sevoflurane induction.

ELIGIBILITY:
Inclusion Criteria:

* Children, 1-9 years old scheduled elective frenectomy under general anesthesia

Exclusion Criteria:

* Patients with an abnormal airway, reactive airway disease, gastroesophageal reflux disease, chronic respiratory disease, or a history of an upper respiratory tract infection in the preceding 6-week period

Ages: 1 Year to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 114 (Actual)
Dates: Start 2012-02; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Intubating condition | Participants will be followed for the duration of intubation, an expected average of 1 minute.
  The investigators will perform the evaluation of intubating condtion through scoring system provided by Viby-Mogensen during intubation procedure. The scoring system is consisted of excellent, good, and poor.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Seoul, South Korea

REFERENCES:
- [Background] Park S, Kim JH, Bae JC, Lee JR, Kim MS. Tracheal intubation with or without a neuromuscular blocking agent for a short surgical procedure in children: Prospective, randomized, double-blind trial. Paediatr Anaesth. 2021 Aug;31(8):863-870. doi: 10.1111/pan.14205. Epub 2021 Jun 3. PMID 33993571